CLINICAL TRIAL: NCT01808001
Title: Critical Event Checklist Use for Management of Critical Events in Ambulatory Surgery
Brief Title: Simulation Team Training and Critical Event Checklist Use for Optimizing the Management of Critical Perioperative Events in an Ambulatory Surgical Facility
Acronym: CEC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0030-B
Record Dates: First submitted 2013-02-27; First posted 2013-03-08 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-02

CONDITIONS: Simulation Team Training in Ambulatory Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will determine if operating room teams manage a simulated event more effectively using a critical event checklist. Performance will be evaluated using a score based on how closely they follow a protocol for critical event management; a 'team' score and a score based on clinical recovery of the simulated patient. All teams will receive a debriefing session after managing 4 scenarios. Teams will return and manage 4 further scenarios after a period of 6-9 months.

The investigators will be testing the hypothesis that both clinical and behavioral team performance will improve with the use of Critical Event Checklists. The investigators also expect that health professional (participant) could attain knowledge related to the importance of non-technical skills and the use of CECs in the management of critical events.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria for Participation:

  1. RN in active practice
  2. Anesthesiologist in active practice
  3. Surgeon in active practice

     Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Health care professionals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
professional health care teams' behavioural performance is measured using a previously validated non-technical skills (NTS) tool (TEAM)and key process checklists | 1.5 years

SECONDARY OUTCOMES:
questionnaires in participants' opinion of the educational intervention, willingness to participate in annual simulated scenario training, effect on subsequent clinical performance and opinion re: best sites for CEC placement | 1.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada